CLINICAL TRIAL: NCT02448303
Title: A Phase 2 Proof-of-Concept Study of the Combination of ACP-196 and Pembrolizumab in Subjects With Advanced Non-small Cell Lung Carcinoma
Brief Title: Pembrolizumab Alone and In Combination With Acalabrutinib (ACP-196) in Subjects With Advanced Non-small Cell Lung Cancer
Acronym: KEYNOTE166
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Acerta Pharma BV (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACE-ST-007
Record Dates: First submitted 2015-05-14; First posted 2015-05-19 (Estimated); Results first posted 2019-09-12 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; acalabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): pembrolizumab
  Interventions: Drug: Pembrolizumab
- Arm 2 (Experimental): acalabrutinib plus pembrolizumab
  Interventions: Drug: Pembrolizumab; Drug: Acalabrutinib

INTERVENTIONS:
Drug: Pembrolizumab
  Other Names: Keytruda
Drug: Acalabrutinib
  Other Names: ACP-196
  Arms: Arm 2

SUMMARY:
Pembrolizumab alone and in combination with acalabrutinib in subjects with advanced non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 years of age
* ECOG performance status of 0 or 1
* Histologically confirmed recurrent or metastatic NSCLC (adenocarcinoma, large cell, squamous cell, or not otherwise specified) that has either progressed during or after platinum-based chemotherapy
* Received at least 1 platinum-based chemotherapy regimen. Note: Subjects with EGFR mutations or ALK translocations are required to have received prior therapy with appropriate TKI; prior platinum-based chemotherapy is not required for this specific patient population

Exclusion Criteria:

* Prior malignancy (other than lung cancer), except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer from which the subject has been disease free for ≥ 2 years or which will not limit survival to < 2 years
* Known central nervous system metastases and/or carcinomatous meningitis
* Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel, symptomatic inflammatory bowel disease, partial or complete bowel obstruction, or gastric restrictions and bariatric surgery, such as gastric bypass
* Breastfeeding or pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Acerta Clinical Trials, Study Director — 1-888-292-9613; acertamc@dlss.com
Locations (1):
- Western Regional Medical Center/Cancer Treatment Center of America, Goodyear, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1 - Pembrolizumab Monotherapy: Pembrolizumab 200mg administered as an intravenous (IV) infusion every 3 weeks (Q3W).
- Arm 2 - Acalabrutinib + Pembrolizumab: Acalabrutinib 100mg PO BID plus Pembrolizumab 200mg administered as an intravenous (IV) infusion every 3 weeks (Q3W).
Period: Overall Study
Arm/Group | Arm 1 - Pembrolizumab Monotherapy | Arm 2 - Acalabrutinib + Pembrolizumab
Started | 38 | 36
Enrolled | 38 | 36
Received Study Medication | 33 | 35
Discontinued Study | 38 | 36
Completed | 0 | 0
Not Completed | 38 | 36

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 - Pembrolizumab Monotherapy | Arm 2 - Acalabrutinib + Pembrolizumab | Total
Number analyzed (Participants) | 33 | 35 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (10.2) | 64.6 (9.33) | 64.2 (9.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 20 | 35
  Male | 18 | 15 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 32 | 34 | 66
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 25 | 27 | 52
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 33 | 35 | 68

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Overall Response
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Every 12 weeks for up to 2 years
Population: The study participants had to have a minimum of one scan (for tumor assessment) after randomization/treatment in order to be considered analyzed.
  And some of the participants didn't make it to Wk 7 of treatment, hence reduction in the number of subjects analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 - Pembrolizumab Monotherapy | Arm 2 - Acalabrutinib + Pembrolizumab
Number analyzed (Participants) | 31 | 28
Participants | 4 | 4

ADVERSE EVENTS:
Time Frame: Safety Analysis tracked from 0 day to 2 years.
Arm/Group | Arm 1 - Pembrolizumab Monotherapy | Arm 2 - Acalabrutinib + Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 18/33 | 23/35
Serious Adverse Events (participants affected / at risk) | 12/33 | 18/35
Other Adverse Events (participants affected / at risk) | 33/33 | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 - Pembrolizumab Monotherapy (N=33) | Arm 2 - Acalabrutinib + Pembrolizumab (N=35)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Large Intestine Haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0 — General Disorders and Administration Site Conditions.
Pain (General disorders) | 0 | 1 — General Disorders and Administration Site Conditions.
Bile Duct Obstructions (Hepatobiliary disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 3
Cellulitis (Infections and infestations) | 0 | 1
Clostridium Difficile Colitis (Infections and infestations) | 0 | 1
Oral Candidiasis (Infections and infestations) | 1 | 0
Pneumonia Viral (Infections and infestations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Failure to Thrive (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Metastases to Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Syncope (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 1
Mental Status Changes (Psychiatric disorders) | 1 | 1
Acute Kidney Injury (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 1
Orthostatic Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 - Pembrolizumab Monotherapy (N=33) | Arm 2 - Acalabrutinib + Pembrolizumab (N=35)
Anaemia (Blood and lymphatic system disorders) | 5 | 9
Ear Pain (Ear and labyrinth disorders) | 2 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 2
Hypothyroidism (Endocrine disorders) | 2 | 2
Diplopia (Eye disorders) | 0 | 2
Diarrhea (Gastrointestinal disorders) | 7 | 11
Nausea (Gastrointestinal disorders) | 5 | 12
Vomiting (Gastrointestinal disorders) | 3 | 13
Constipation (Gastrointestinal disorders) | 3 | 7
Dry Mouth (Gastrointestinal disorders) | 3 | 5
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 4
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 2 | 2
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 3
Oesophagitis (Gastrointestinal disorders) | 1 | 2
Stomatitis (Gastrointestinal disorders) | 1 | 2
Fatigue (General disorders) | 15 | 9 — General Disorders & Administration Site Conditions.
Oedema Peripheral (General disorders) | 5 | 7 — General Disorders & Administration Site Conditions.
Pyrexia (General disorders) | 3 | 4 — General Disorders & Administration Site Conditions.
Non-Cardiac Chest Pain (General disorders) | 1 | 5 — General Disorders & Administration Site Conditions.
Asthenia (General disorders) | 0 | 2 — General Disorders & Administration Site Conditions.
Chest Pain (General disorders) | 2 | 0 — General Disorders & Administration Site Conditions.
Seasonal Allergy (Immune system disorders) | 2 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 5
Pneumonia (Infections and infestations) | 2 | 2
Urinary Tract Infection (Infections and infestations) | 2 | 2
Oral Candidiasis (Infections and infestations) | 2 | 2
Bronchitis (Infections and infestations) | 2 | 1
Nasopharyngitis (Infections and infestations) | 3 | 0
Chills (General disorders) | 1 | 3 — General Disorders & Administration Site Conditions.
Mucosal Inflammation (General disorders) | 2 | 0 — General Disorders & Administration Site Conditions.
Pain (General disorders) | 1 | 2 — General Disorders & Administration Site Conditions.
Sinusitis (Infections and infestations) | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 3
Aspartate Aminotransferase Increased (Investigations) | 2 | 5
Weight Decreased (Investigations) | 3 | 5
Blood Creatinine Increased (Investigations) | 2 | 4
Alanine Aminotransferase Increased (Investigations) | 0 | 3
Electrocardiogram QT Prolonged (Investigations) | 1 | 3
Lymphocyte Count Decreased (Investigations) | 1 | 2
Amylase Increased (Investigations) | 2 | 0
Weight Increased (Investigations) | 2 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 6 | 12
Dehydration (Metabolism and nutrition disorders) | 6 | 6
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 7
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 4
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 3 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 3
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 | 3
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 3
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Dizziness (Nervous system disorders) | 4 | 7
Headache (Nervous system disorders) | 6 | 6
Dysgeusia (Nervous system disorders) | 2 | 2
Neuropathy Peripheral (Nervous system disorders) | 3 | 1
Somnolence (Nervous system disorders) | 1 | 2
Anxiety (Psychiatric disorders) | 2 | 4
Depression (Psychiatric disorders) | 2 | 3
Insomnia (Psychiatric disorders) | 1 | 3
Confusional State (Psychiatric disorders) | 1 | 2
Sleep Disorder (Psychiatric disorders) | 0 | 2
Acute Kidney Injury (Renal and urinary disorders) | 2 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 10
Wheezing (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Upper-Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 5 | 3
Dry Skin (Skin and subcutaneous tissue disorders) | 2 | 3
Rash Maculo-Papular (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Decubitus Ulcer (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Petechiae (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Hypotension (Vascular disorders) | 2 | 5
Hypertension (Vascular disorders) | 2 | 4
Hot Flush (Vascular disorders) | 2 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 | 4
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1 | 2
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 3
Purpura (Skin and subcutaneous tissue disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-05-23): https://cdn.clinicaltrials.gov/large-docs/03/NCT02448303/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-30): https://cdn.clinicaltrials.gov/large-docs/03/NCT02448303/SAP_001.pdf